CLINICAL TRIAL: NCT02476084
Title: Biomarker Signature and Musculoskeletal Ultrasound Profile in Rheumatoid Arthritis Patients: a Pilot Observational Study
Brief Title: Biomarker Signature and Musculoskeletal Ultrasound Profile in Rheumatoid Arthritis Patients
Acronym: BMUS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 149600
Record Dates: First submitted 2015-05-19; First posted 2015-06-19 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and and Biologic samples collected will be processed in the CTU Translational Research Lab and stored within the Botnar Research Centre adhering to local guidelines on sample requirements, handling and storage. All biological samples will be available for future studies for biomarker profiling.
  The following blood samples will be drawn in order:
  1. Two (10.0ml) K2EDTA tube
  2. One (5.0ml) SST tube
  3. One (3 ml) Tempus RNA tube
  4. One (6 ml) DNA EDTA tube (only during Visit 1)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Conventional synthetic DMARD naïve: Naive RA patients commencing Methotrexate and Hydroxychloroquine.
  Musculoskeletal Ultrasound imaging, synovial biopsy, biological samples collection, questionnaires.
  Interventions: Other: Musculoskeletal Ultrasound Imaging; Other: Synovial biopsy; Other: Biological samples collection; Other: Questionnaires
- DMARD-IR: anti-TNF: Conventional synthetic DMARD inadequate responders commencing Anti-TNF
  Musculoskeletal Ultrasound imaging, synovial biopsy, biological samples collection, questionnaires.
  Interventions: Other: Musculoskeletal Ultrasound Imaging; Other: Synovial biopsy; Other: Biological samples collection; Other: Questionnaires
- DMARD-IR: anti-IL6: Conventional synthetic DMARD inadequate responders commencing anti-IL6
  Musculoskeletal Ultrasound imaging, synovial biopsy, biological samples collection, questionnaires.
  Interventions: Other: Musculoskeletal Ultrasound Imaging; Other: Synovial biopsy; Other: Biological samples collection; Other: Questionnaires
- DMARD-IR: anti-CTLA-4: Conventional synthetic DMARD inadequate responders commencing anti-CTLA-4
  Musculoskeletal Ultrasound imaging, synovial biopsy, biological samples collection, questionnaires.
  Interventions: Other: Musculoskeletal Ultrasound Imaging; Other: Synovial biopsy; Other: Biological samples collection; Other: Questionnaires
- DMARD-IR: anti-CD20: Conventional synthetic DMARD inadequate responders commencing anti-CD20
  Musculoskeletal Ultrasound imaging, synovial biopsy, biological samples collection, questionnaires.
  Interventions: Other: Musculoskeletal Ultrasound Imaging; Other: Synovial biopsy; Other: Biological samples collection; Other: Questionnaires

INTERVENTIONS:
Other: Musculoskeletal Ultrasound Imaging — B-mode and PD musculoskeletal ultrasound examination of selected joints.
Other: Synovial biopsy — US guided synovial biopsy of an inflamed joint including wrists, MCP joints and knees.
Other: Biological samples collection — Draw of research blood samples.
Other: Questionnaires — Administration of validated patients' questionnaires.

SUMMARY:
The purpose of this study is to determine the kinetics of change in quantitative measures of joint inflammation by state of the art power Doppler vascular imaging and to identify biomarkers in biological samples (synovial biopsies, DNA, RNA, PBMC, serum, plasma, urine and stool samples) from parallel cohorts of RA patients undergoing different treatments. This will be achieved implementing MSUS assessments, standard laboratories techniques (such as ELISAs, gene profiling, transcriptome analysis etc.) and the novel CyTOF™ technology.

ELIGIBILITY:
Inclusion Criteria:

* Written confirmed diagnosis of Rheumatoid Arthritis as per ACR/EULAR 2010 criteria.
* If patient is on oral corticosteroids, dose must be stable for 6 weeks prior to baseline visit.
* Willingness and ability to comply with all the study procedures.

Exclusion Criteria:

* Any systemic inflammation conditions (other than RA), connective tissue disease or chronic pain disorders that may interfere with the interpretation of the outcome data. Examples include psoriatic arthritis, reactive arthritis, gout, systemic lupus erythematosus (SLE), polymyalgia rheumatic and/or temporal arteritis, Lyme's disease, fibromyalgia and chronic fatigue syndromes.
* Major surgery planned within 8 weeks prior to screening or planned surgery throughout the study period.
* Treatment with any investigational agent ≤ 4 weeks prior to baseline (or 5 ≤ half-lives of the investigational drug, whichever is the longer).
* Intramuscular/intra-articular glucocorticoids for 6 weeks prior to baseline visit.
* Active infection.
* Septic arthritis within a native joint within the last 12 months.
* Sepsis of a prosthetic joint within 12 months or indefinitely if the joint remains in situ.
* Known HIV or hepatitis B/C infection.
* Latent TB infection unless they have completed adequate antibiotic prophylaxis.
* Malignancy (other than basal cell carcinoma) within the last 10 years.
* New York Heart Association (NYHA) grade 3 or 4 congestive cardiac failure.
* Demyelinating disease.
* Presence of a transplanted organ (with the exception of a corneal transplant > 3 months prior to screening).
* Known recent substance abuse (drug or alcohol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis Patients
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in synovial thickness and vascularity using a limited joint set musculoskeletal ultrasound examination in Rheumatoid Arthritis. | 3 years

SECONDARY OUTCOMES:
Changes in the distribution of cell populations in biological samples from Rheumatoid Arthritis patients using CyTOF. | 3 years
Changes in gene expression in biological samples from Rheumatoid Arthritis patients using gene profiling. | 3 years
Changes in cytokines' concentration in biological samples from Rheumatoid Arthritis patients using ELISA and transcriptome analysis. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Taylor, PhD, FRCP, Principal Investigator — Kennedy Institute of Rheumatology, University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, United Kingdom